CLINICAL TRIAL: NCT02744742
Title: Granulocyte Colony-stimulating Factor+Decitabine+Busulfan+Cyclophosphamide vs Busulfan+Cyclophosphamide Conditioning Regimen for Patients With RAEB-1, RAEB-2 and AML Secondary to MDS Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: G-CSF+Decitabine+BUCY vs BUCY Conditioning Regimen for RAEB-1, REAB-2 and AML Secondary to MDS Undergoing Allo-HSCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Institute of Hematology & Blood Diseases Hospital, China (Other); Peking University People's Hospital (Other); First People's Hospital of Chenzhou (Other); Liuzhou Workers' Hospital (Other Government)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-CSF+Dec+BUCYvsBUCY-MDS-2016
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2016-04

CONDITIONS: Myelodysplastic Syndrome; Allogeneic Hematopoietic Stem Cell Transplantation; Conditioning
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine; Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF + Decitabine + BUCY (Experimental): For patients with RAEB-1, REAB-2 and AML Secondary to MDS undergoing allo-HSCT ，Granulocyte Colony-Stimulating Factor(G-CSF)+Decitabine+BUCY conditioning regimen was G-CSF 5-10ug/kg/day on days -17 and -10 (when white blood cell is more than 20G/L, stop using G-CSF)；Decitabine 20mg/m2/day on days -14 and -10； Busulfan (BU) 3.2 mg/kg/day on days -7 and -4；Cyclophosphamide (CY) 60 mg/kg/day on days -3 and -2.
  Interventions: Drug: Decitabine; Drug: Busulfan (BU); Drug: Cyclophosphamide (CY); Drug: Granulocyte Colony-Stimulating Factor(G-CSF)
- BUCY (Active Comparator): For patients with RAEB-1, REAB-2 and AML Secondary to MDS undergoing allo-HSCT ，BUCY conditioning regimen was Busulfan (BU) 3.2 mg/kg/day on days -7 and -4；Cyclophosphamide (CY) 60 mg/kg/day on days -3 and -2.
  Interventions: Drug: Busulfan (BU); Drug: Cyclophosphamide (CY)

INTERVENTIONS:
Drug: Decitabine — Decitabine was administered at 20mg/m2/day on days -14 and -10.
  Arms: G-CSF + Decitabine + BUCY
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days -7 to -4.
Drug: Cyclophosphamide (CY) — Cyclophosphamide was administered at 60 mg/kg/day on days -3 to -2.
Drug: Granulocyte Colony-Stimulating Factor(G-CSF) — G-CSF was administered at 5-10 ug/kg/day on days -17 and -10. When white blood cell is more than 20G/L, stop using G-CSF.
  Arms: G-CSF + Decitabine + BUCY

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) appears to be an efficient tool to cure refractory anemia with excess blasts-1 (RAEB-1), refractory anemia with excess blasts-2 (RAEB-2) and acute myeloid leukemia (AML) secondary to myelodysplastic syndrome (MDS). At present, the best conditioning regimen for RAEB-1, RAEB-2 and AML secondary to MDS undergoing allo-HSCT remains in discussion. In this prospective randomized controlled study, the safety and efficacy of G-CSF+ Decitabine + BUCY and BUCY myeloablative conditioning regimens in patients with RAEB-1, REAB-2 and AML Secondary to MDS undergoing allo-HSCT are evaluated.

DETAILED DESCRIPTION:
Allo-HSCT appears to be an efficient tool to cure patients with MDS and AML secondary to MDS. At present, the best conditioning regimen for MDS and AML secondary to MDS undergoing allo-HSCT remains in discussion. BUCY conditioning regimen is the standard myeloablative regimen for MDS and AML secondary to MDS undergoing allo-HSCT. However, it appears to have higher relapse rate. To reduce the relapse rate, decitabine is added in the conditioning regimen. In this prospective randomized controlled study, the safety and efficacy of G-CSF + Decitabine + BUCY and BUCY myeloablative conditioning regimens in RAEB-1, REAB-2 and AML secondary to MDS undergoing allo-HSCT are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* RAEB-1, REAB-2 and AML Secondary to MDS undergoing allo-HSCT
* 14-65 years

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
relapse rate | 2 year

SECONDARY OUTCOMES:
overall survival (OS) | 2 year
disease-free survival (DFS) | 2 year
transplant-related mortality (TRM) | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Xuan L, Dai M, Jiang E, Wang Y, Huang F, Fan Z, Xu N, Nie D, Liang X, Chen H, Ye J, Shi P, Liu H, Jin H, Lin R, Yan C, Zhang Y, Sun J, Han M, Liu Q. The effect of granulocyte-colony stimulating factor, decitabine, and busulfan-cyclophosphamide versus busulfan-cyclophosphamide conditioning on relapse in patients with myelodysplastic syndrome or secondary acute myeloid leukaemia evolving from myelodysplastic syndrome undergoing allogeneic haematopoietic stem-cell transplantation: an open-label, multicentre, randomised, phase 3 trial. Lancet Haematol. 2023 Mar;10(3):e178-e190. doi: 10.1016/S2352-3026(22)00375-1. Epub 2023 Jan 23. PMID 36702138